CLINICAL TRIAL: NCT03195725
Title: How is the Term 'Harm' Being Interpreted and Documented on Hospice DNACPR Forms Following the Tracey Judgement?
Status: Completed | Type: Observational
Sponsor: The Royal Wolverhampton Hospitals NHS Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2017PAL94
Record Dates: First submitted 2017-06-20; First posted 2017-06-22 (Actual); Last update posted 2019-06-19 (Actual); Status verified 2019-06

CONDITIONS: Cardiopulmonary Resuscitation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Year 2013: Participant's notes will be reviewed from the year 2013
  Interventions: Other: Review of notes
- Year 2015: Participant's notes will be reviewed from the year 2015
  Interventions: Other: Review of notes

INTERVENTIONS:
Other: Review of notes — No intervention will occur

SUMMARY:
To investigate how discussions surrounding Do Not Attempt Cardiopulmonary Resuscitation (DNACPR) decisions have changed following the Tracey judgement and how "harm" is being defined by clinicians working within specialist palliative care in a hospice setting.

DETAILED DESCRIPTION:
This is a retrospective case note review. Five hospices within the West Midlands will be invited to participate and up to 300 sets of deceased patients' notes containing a DNACPR form will be reviewed; 150 from 2013 (prior to the Tracey judgement) and 150 from 2015 (following the Tracey judgement).

Initially these forms will be reviewed to document the percentage of patients with whom a DNACPR decision was discussed in 2013 and the percentage with whom it was discussed in 2015 to allow comparison from before the Tracey judgement and after the Tracey judgement.

If patients did NOT have DNACPR decisions discussed with them, their DNACPR forms and clinical notes will then be reviewed and the reasons documented for not involving patients in 2013 and in 2015 compared. It is anticipated that many, if not most, DNACPR decisions which were not discussed with patients in 2013 will cite "distress" as the reason but following the Tracey judgement this would not be acceptable in 2015.

Further analysis of DNACPR forms and clinical notes will then take place for those patients identified as not being involved in DNACPR discussions in 2015 (post-Tracey) to identify whether, and how, "harm" was defined by the clinician. This should be recorded on the DNACPR form or in the clinical notes.

Following data collection, quantitative analysis will be undertaken to allow comparison of percentages of DNACPR decisions discussed with patients in 2013 and 2015 followed by descriptive analysis of variation in reasons for not discussing DNACPR decisions in 2013 and 2015. This study is explorative in nature and further qualitative analysis will not be part of this research project.

ELIGIBILITY:
Inclusion Criteria:

* Patients who died in 2013 or 2015 known to the individual hospice team (in-patient unit, day unit or community team)
* Completed DNACPR form within the clinical notes which was completed in 2013 or 2015

Exclusion Criteria:

* No completed DNACPR form within the clinical notes
* DNACPR form not completed in 2013 or 2015

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Deceased patients' notes will be reviewed from 2013 (prior to the Tracey judgement) and from 2015 (following the Tracey judgement).
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2017-07-24 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2018-10-31 (Actual)

PRIMARY OUTCOMES:
The number of DNACPR decisions | 1 year
  1) The number of DNACPR decisions which were discussed with patients in 2013 (prior to the Tracey judgement) and in 2015 (following the Tracey judgement)
The reasons for not discussing DNACPR decisions | 1 year
  2) The reasons documented on DNACPR forms and in clinical notes for not discussing DNACPR decisions in 2013 and in 2015

SECONDARY OUTCOMES:
The documentation of the concept of 'harm' in DNACPR decisions | 1 year
  The documentation of the concept of 'harm' in DNACPR decisions not discussed with patients in 2015

CONTACTS AND LOCATIONS:
Locations (1):
- Compton Hospice, Wolverhampton, United Kingdom

IPD SHARING:
Plan to Share IPD: No